CLINICAL TRIAL: NCT06932614
Title: Comparing the Efficacy of Lyophilized Self Growth Factor Versus Platelet-Rich Plasma(PRP) Injection for Knee Osteoarthritis: A Prospective, Double-Blind, Randomized Controlled Trial
Brief Title: Comparing the Efficacy of Lyophilized Self Growth Factor Versus PRP Injection for Knee OA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Yu-CHI Su, Attending Physician and lecturer of Department of Physical Medicine and Rehabilitation, Tri-Service General Hospital
Allocation: Not Applicable | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C202404004
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis; PRP Injection
Keywords: Knee Osteoarthritis; PRP injection
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lyophilized self growth factor (Experimental): Knee Intraarticular injection with Lyophilized self growth factor
  Interventions: Procedure: Lyophilized self growth factor
- Platelet-Rich Plasma(PRP) (Active Comparator): Knee intraarticular injection with Platelet-Rich Plasma(PRP)
  Interventions: Procedure: Platelet-Rich Plasma(PRP)
- normal saline (Placebo Comparator): Knee intraarticular injection with normal saline
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Lyophilized self growth factor — Knee Intraarticular injection with Lyophilized self growth factor
  Arms: Lyophilized self growth factor
Procedure: Platelet-Rich Plasma(PRP) — Knee Intraarticular injection with Lyophilized self growth factor
  Arms: Platelet-Rich Plasma(PRP)
Procedure: Placebo — Knee Intraarticular injection with normal saline
  Arms: normal saline

SUMMARY:
Knee osteoarthritis(OA) is a common degenerative joint disease that often leads to knee pain, stiffness, and a decline in quality of life among middle-aged and elderly individuals. Platelet-rich plasma (PRP) is a regenerative treatment method that involves drawing a small amount of the patient's own blood and using centrifugation process to produce PRP. PRP, which is rich in growth factors and anti-inflammatory cytokines, facilitate the repair of damaged tissues and has been used in treating knee OA. Self-repair factor (SRF), an advanced form of PRP, is created using multi-step centrifugation and proprietary processes to increase platelet concentration. This enhancement may offer superior repair efficacy and faster recovery compared to traditional PRP. To explore this potential, we designed a randomized, double-blind, clinical trial to compare the effectiveness of SRF and PRP in treating degenerative knee osteoarthritis.

DETAILED DESCRIPTION:
Knee osteoarthritis(OA) is a common degenerative joint disease that often leads to knee pain, stiffness, and a decline in quality of life among middle-aged and elderly individuals. Treatment options include weight loss, anti-inflammatory and pain-relieving medications, physical rehabilitation, and intra-articular injections of corticosteroids or hyaluronic acid. However, these methods often have limited efficacy or may cause side effects. Platelet-rich plasma (PRP) is a regenerative treatment method that involves drawing a small amount of the patient's own blood and using centrifugation process to produce PRP. PRP, which is rich in growth factors and anti-inflammatory cytokines, facilitate the repair of damaged tissues and has been used in treating knee OA. However, there is still lack of strong evidence of the therapeutic effects of PRP injection in knee OA. Therefore, there is a need to investigate novel therapies for knee OA. Self-repair factor (SRF), an advanced form of PRP, is created using multi-step centrifugation and proprietary processes to increase platelet concentration. This enhancement may offer superior repair efficacy and faster recovery compared to traditional PRP. To explore this potential, we designed a randomized, double-blind, clinical trial to compare the effectiveness of SRF and PRP in treating degenerative knee osteoarthritis. Patients with mild to moderate knee osteoarthritis who have experienced symptoms for more than three months. 30 participants will be recruited and randomly divided into three groups: the SRF group, the PRP group, and a control group. Each participant will receive knee intra-articular injections as part of a three-month treatment regimen, with one injection per month for a total of three injections. Patients will be evaluated before the trial, and at one, two, three, and six months after the injections. Clinical outcomes will be assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), the Intermittent and Constant Osteoarthritis Pain (ICOAP) scale, the sit-to-stand test, and the Visual Analog Scale (VAS) for pain. The study aims to confirm the clinical efficacy of SRF in treating degenerative knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged over 20 and under 80.
* Consciousness clear and able to communicate.
* Unilateral or bilateral osteoarthritis of the knee with symptoms lasting more than 3 months.
* X-ray imaging shows mild to moderate knee osteoarthritis (Kellgren-Lawrence grades 1-3).
* Knee joint pain with a Visual Analogue Scale (VAS) score greater than 4.

Exclusion Criteria:

* Severe knee osteoarthritis (Kellgren-Lawrence grade 4).
* Currently systemic infection.
* Received hyaluronic acid or corticosteroid intraarticular injections within the past six months, or received NSAIDs or oral corticosteroid treatment within 7 days prior to treatment.
* The treated joint has undergone joint replacement surgery or major surgery.
* Severe knee deformity or instability.
* Known history of cancers, rheumatoid arthritis, platelet dysfunction, thrombocytopenia, hypofibrinogenemia, acute or chronic infectious diseases, chronic liver disease, or poorly controlled cardiovascular disease or diabetes.
* Currently receiving anticoagulant therapy.
* Long-term or excessive use of aspirin or vitamin E.
* History of HIV/AIDS, syphilis, or other legally notifiable infectious diseases.
* Pregnant or breastfeeding women, or women and men of childbearing potential who are unable to use effective contraception during the treatment period.
* Deemed unsuitable for participation in the trial by the principal investigator.
* Unable to sign the informed consent form.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index | Pre-treatment, 1st month, 2nd month, 3rd month, 6th month
  The structure and function of the knee joint are assessed from three main aspects: pain, stiffness, and joint function, with a total of 24 items. The pain section consists of 5 items (24 points in total), the stiffness section has 2 items (8 points in total), and the joint function section includes 17 items (68 points in total). A lower score indicates more severe pain, stiffness, and a higher degree of disability.

SECONDARY OUTCOMES:
Visual Analogue Scale | Pre-treatment, 1st month, 2nd month, 3rd month, 6th month
  Change from baseline of pain on 1st month, 2nd month, 3rd month, 6th month after injection.
  Pain severity was evaluated using visual analog scale (VAS). Pain score scale ranged from 0 to 10, with 10 indicating the most severe pain
The intermittent and constant pain score , ICOAP | Pre-treatment, 1st month, 2nd month, 3rd month, 6th month
  The content is divided into two subcategories: continuous pain (5 items) and intermittent pain (6 items), with a total of 11 items. Each item is scored from 0, representing no pain, to 4, representing extreme pain. A higher score indicates more severe pain. The Chinese version has reliable validity and reliability.
Timed Up and Go test | Pre-treatment, 1st month, 2nd month, 3rd month, 6th month.
  Align the chair legs with the starting baseline and place a cone 3 meters ahead. The participant sits in the chair with their feet naturally bent, stands up comfortably, walks forward for 3 meters, turns around, and walks back to sit down. The time taken to complete the task is recorded. This test has good validity and reliability for assessing the mobility of patients with degenerative knee osteoarthritis.

CONTACTS AND LOCATIONS:
Locations (1):
- No. 325, Sec. 2, Chenggong Rd., Neihu Dist., Taipei, Taiwan

REFERENCES:
- [Background] Woodell-May J, Matuska A, Oyster M, Welch Z, O'Shaughnessey K, Hoeppner J. Autologous protein solution inhibits MMP-13 production by IL-1beta and TNFalpha-stimulated human articular chondrocytes. J Orthop Res. 2011 Sep;29(9):1320-6. doi: 10.1002/jor.21384. Epub 2011 Mar 15. PMID 21437966
- [Background] Jo CH, Kim JE, Yoon KS, Shin S. Platelet-rich plasma stimulates cell proliferation and enhances matrix gene expression and synthesis in tenocytes from human rotator cuff tendons with degenerative tears. Am J Sports Med. 2012 May;40(5):1035-45. doi: 10.1177/0363546512437525. Epub 2012 Feb 23. PMID 22366517
- [Background] Chavda S, Rabbani SA, Wadhwa T. Role and Effectiveness of Intra-articular Injection of Hyaluronic Acid in the Treatment of Knee Osteoarthritis: A Systematic Review. Cureus. 2022 Apr 26;14(4):e24503. doi: 10.7759/cureus.24503. eCollection 2022 Apr. PMID 35651409
- [Background] Arroll B, Goodyear-Smith F. Corticosteroid injections for osteoarthritis of the knee: meta-analysis. BMJ. 2004 Apr 10;328(7444):869. doi: 10.1136/bmj.38039.573970.7C. Epub 2004 Mar 23. PMID 15039276
- [Background] Loeser RF, Goldring SR, Scanzello CR, Goldring MB. Osteoarthritis: a disease of the joint as an organ. Arthritis Rheum. 2012 Jun;64(6):1697-707. doi: 10.1002/art.34453. Epub 2012 Mar 5. No abstract available. PMID 22392533
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Neogi T. The epidemiology and impact of pain in osteoarthritis. Osteoarthritis Cartilage. 2013 Sep;21(9):1145-53. doi: 10.1016/j.joca.2013.03.018. PMID 23973124